CLINICAL TRIAL: NCT03135743
Title: Retrospective Analysis of Lymphomas and Cancers Synchronous Occurrence in Picardy From 2007 to 2012
Acronym: LYMPHOSYNCHRO
Status: Withdrawn | Type: Observational
Why Stopped: No patients enrolled
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2016_843_0024
Record Dates: First submitted 2017-04-27; First posted 2017-05-01 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma; Cancer
MeSH Terms: conditions — Lymphoma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Show an increase in incidence of cancers in patients with synchronous lymphoma — Show an increase in incidence of cancers in patients with synchronous lymphoma

SUMMARY:
Cancer is the leading cause of death in man and the second leading cause in women with 85,000 and 63,000 deaths, respectively, in 2012. A working group led by Holly L. Howe, PhD, in 2002 defined primary neoplasia Such as the occurrence and diagnosis of two or more independent neoplasms of different histology in the same patient. The occurrence of a new cancer has become more frequent in recent years: the prevalence of multiple primary neoplasia (NPM) is estimated between 0.73% and 11.7%. According to the French data, the risk of second cancer in people who have already had a first cancer is increased by 36% compared to the general population. Several studies have reported an increase in the risk of cancer after treatment of lymphoma but there are currently no studies on the occurrence of lymphoma and cancer of synchronous occurrence.

In our department, 19 patients presented cancer and lymphoma synchronously, that is to say 6 months between 2007 and 2012.

The main objective is to show that there is an increase in the incidence of cancers in patients diagnosed for lymphoma synchronously. Secondary objectives are to describe the clinical and biological characteristics of the patients concerned and to formulate hypotheses on the physiopathological mechanisms involved: peri-tumoral B-cell lymphoproliferation, alteration of the immune system or rearrangement of the BCR.

In a second step, the investigator could propose a multicenter epidemiological study using data from the different Cancer Registries. If results are confirmed in a larger cohort, recommendations could be made.

ELIGIBILITY:
Inclusion Criteria:

* Being older than 18
* Have been diagnosed for Hodgkin's or non-Hodgkin's lymphoma from 1 January 2007 to 31 December 2012
* Diagnostic confirmation either in anatomopathology or in cytology
* Delay of 6 months maximum between the two neoplasms (Synchronic / metachronous distinction)

Exclusion Criteria:

* Hemopathy other than lymphoma (CLL and lymphocytic lymphoma excluded)
* Diagnosis of lymphoma outside the inclusion period Metastases and recurrences were not considered as secondary cancers, but as relapses of the first neoplasia
* Cutaneous squamous cell carcinomas were not considered secondary cancer because of the absence of available incidence data (FRANCIM network)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective study on data and elements of the human body (anatomo-pathological blade) over a period of 6 years in patients with synchronous lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-08-20 (Estimated); Primary Completion 2019-06-20 (Estimated); Study Completion 2019-06-20 (Estimated)

PRIMARY OUTCOMES:
Analysis of the occurrence of cancer and lymphoma within 6 months between 2007 and 2012 | 5 years